CLINICAL TRIAL: NCT01797653
Title: The Effects of CPAP-withdrawal on Microvascular Function in Patients With Obstructive Sleep Apnea: A Randomized-controlled Trial
Brief Title: Randomized-controlled Trial (RCT) on CPAP-withdrawal and Microvascular Function in OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPAP_V1.0 (01.11.2012)
Record Dates: First submitted 2013-02-15; First posted 2013-02-22 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Obstructive Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo CPAP (Placebo Comparator): patients established on CPAP therapy, who are randomized to the placebo comparator, will use a CPAP device with subtherapeutic pressure during two weeks.
  Interventions: Other: CPAP therapy withdrawal
- therapeutic CPAP (Active Comparator): patients who are randomized to the active comparator, will continue with CPAP treatment with therapeutic pressure during two weeks
  Interventions: Procedure: Continue CPAP treatment

INTERVENTIONS:
Other: CPAP therapy withdrawal — CPAP (continuous positive airway pressure) with subtherapeutic pressure during two weeks
  Other Names: CPAP treatment with subtherapeutic pressure
  Arms: Placebo CPAP
Procedure: Continue CPAP treatment — Continue treatment with therapeutic continuous positive airway pressure device
  Other Names: therapeutic continuous positive airway pressure device
  Arms: therapeutic CPAP

SUMMARY:
Randomized controlled trial (therapeutic vs. placebo CPAP) including 46 patients with obstructive sleep apnea (OSA) to define the physiological effects of continuous positive airway pressure (CPAP) therapy withdrawal on myocardial perfusion and dermal and renal microvascular function during a 2 week period.

ELIGIBILITY:
Inclusion criteria:

* Objectively confirmed OSA (at the time of original diagnosis) with an oxygen desaturation index (ODI, =4% dips) of >20/h and an ESS of >10.
* Currently >20/h oxygen desaturations (=4% dips) during an ambulatory nocturnal pulse oximetry performed at the end of a 4-night period without CPAP.
* Treated with CPAP for more than 12 months, minimum compliance 4h per night, AHI<10 with treatment (according to CPAP machine download data).
* Current ESS <10.

Exclusion criteria:

* Previous ventilatory failure (awake SpO2 <93% and PaCO2>6kPa).
* Unstable, untreated coronary or peripheral artery disease, severe arterial hypertension or hypotension (>180/110 or <90/60mmHg)
* Previously diagnosed with Cheyne-Stokes breathing.
* Current professional driver; Any previous sleep related accident.
* Age <20 or >75 years at trial entry.
* Acute inflammatory disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
hyperaemic myocardial blood flow | 2 weeks

SECONDARY OUTCOMES:
Coronary flow reserve | 2 weeks
  Coronary flow reserve determined by PET
Urine albumine excretion rate | 2 weeks
Dermal microvascular vasodilatory response | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof MD, Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Schwarz EI, Furian M, Schlatzer C, Stradling JR, Kohler M, Bloch KE. Nocturnal cerebral hypoxia in obstructive sleep apnoea: a randomised controlled trial. Eur Respir J. 2018 May 30;51(5):1800032. doi: 10.1183/13993003.00032-2018. Print 2018 May. PMID 29700104
- [Derived] Turnbull CD, Rossi VA, Santer P, Schwarz EI, Stradling JR, Petousi N, Kohler M. Effect of OSA on hypoxic and inflammatory markers during CPAP withdrawal: Further evidence from three randomized control trials. Respirology. 2017 May;22(4):793-799. doi: 10.1111/resp.12946. Epub 2016 Nov 18. PMID 27860068
- [Derived] Schwarz EI, Schlatzer C, Rossi VA, Stradling JR, Kohler M. Effect of CPAP Withdrawal on BP in OSA: Data from Three Randomized Controlled Trials. Chest. 2016 Dec;150(6):1202-1210. doi: 10.1016/j.chest.2016.07.012. Epub 2016 Jul 21. PMID 27452767
- [Derived] Stradling JR, Schwarz EI, Schlatzer C, Manuel AR, Lee R, Antoniades C, Kohler M. Biomarkers of oxidative stress following continuous positive airway pressure withdrawal: data from two randomised trials. Eur Respir J. 2015 Oct;46(4):1065-71. doi: 10.1183/09031936.00023215. Epub 2015 May 28. PMID 26022961